CLINICAL TRIAL: NCT04967261
Title: The Evaluation of Optimal Observation Period for Neurological Recovery in Post-arrest Survivors
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106019RINB
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2021-07

CONDITIONS: Cardiology
Keywords: Cardiac arrest; post-cardiac arrest syndrome; neurological outcome
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore whether the patient's neurological function recovery period is sufficient after successful emergency resuscitation recommended by the current guidelines

DETAILED DESCRIPTION:
The research team will collect patient data after successful emergency resuscitation after cardiac arrest in the emergency room of National Taiwan University Hospital, and will collect and analyze the relationship between the time for patients to regain consciousness and drug use, hemodynamic changes, and neurological examination results after resuscitation. To explore whether the patient population needs to extend the observation time of neurological function after a certain CPR emergency treatment, and allow the patient to have a longer observation period to regain consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-traumatic cardiac arrest in the emergency room of National Taiwan University Hospital (including pre-hospital cardiac arrest and in-hospital cardiac arrest) after successful emergency resuscitation

Exclusion Criteria:

* Under 20 years old
* Pregnant women
* Those who have not been admitted to the intensive care unit
* Unconsciousness before the heartbeat stops
* A clear consciousness after successful first aid resuscitation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-traumatic cardiac arrest who have been successfully resuscitated by first aid and admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongshan South Road, Taiwan